CLINICAL TRIAL: NCT00861393
Title: The Impact of a Brief Cognitive Behavior Therapy Intervention Aimed at Improving Emotional Well-Being and Quality of Life for Individuals With Spinal Cord Injuries
Brief Title: Cognitive Behavioural Therapy (CBT) For Improving Emotional Well Being in Spinal Cord Injuries (SCI)
Acronym: CBT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Toronto Rehabilitation Institute (Other)
Responsible Party: Dr. Cheryl Bradbury, C.Psych, Toronto Rehabilitation Institute
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CBT-08-06
Record Dates: First submitted 2009-03-12; First posted 2009-03-13 (Estimated); Last update posted 2009-03-13 (Estimated); Status verified 2009-03

CONDITIONS: Spinal Cord Injuries
MeSH Terms: conditions — Spinal Cord Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- CBT (Other)
  Interventions: Behavioral: CBT
- Waitlist (Other)
  Interventions: Behavioral: Waitlist CBT

INTERVENTIONS:
Behavioral: CBT — 12 Session CBT group
  Arms: CBT
Behavioral: Waitlist CBT — Participants in the waitlist will receive CBT when first group has completed CBT and been tested.
  Arms: Waitlist

SUMMARY:
The purpose of the study is to determine whether or not a brief psychological treatment called cognitive behaviour therapy will help people who have suffered a spinal cord injury to cope better with their current circumstances.

DETAILED DESCRIPTION:
The goal of the current proposed research project is to investigate the potential efficacy of a group cognitive behavioural therapy (CBT) intervention aimed at improving emotional well-being, specifically mood, adjustment and quality of life (QOL), after Spinal Cord Injury(SCI). The intervention will be adapted to meet the unique needs of patients suffering from an SCI. The study objectives are:

(1) to evaluate the impact of a brief CBT intervention aimed at decreasing emotional distress and improving quality of life; (2) to evaluate the sustainability of CBT therapeutic gains over time; (3) to conduct sub group analyses in order to better determine why some patients may improve post CBT, while others may not.

ELIGIBILITY:
Inclusion Criteria:

* between ages 18-65
* diagnosed with spinal cord injury
* currently endorsing significant distress as measured
* able to provide informed consent
* if taking psychoactive meds, on a stable dosage
* are not currently enrolled in any other psychological treatment program
* speak basic english with no diagnosis of communication disorder

Exclusion Criteria:

* they endorse current suicidal ideation
* have a Neurodegenerative disorder such as Multiple Sclerosis

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2009-02; Primary Completion 2010-01 (Estimated); Study Completion 2010-01 (Estimated)

PRIMARY OUTCOMES:
Symptom checklist -90-R (SCL-90-R) Depression Anxiety Stress Scales (DASS-21) Personality Assessment Inventory (PAI) PAI measure a broad range of psychological symptoms and personality characteristics. | one year

SECONDARY OUTCOMES:
The Ways of Coping Scale- Revised (WOC-R) Community Integration Questionnaire (CIQ) Satisfaction with Life Scale (SWLS) Life satisfaction Checklist (LiSat-11) Stage of change Scales (SOC) | one year

CONTACTS AND LOCATIONS:
Locations (1):
- Toronto Rehabilitation Institute (Lyndhurst Center), Toronto, Ontario, Canada